CLINICAL TRIAL: NCT05981456
Title: The Effect of Flipped Education Model on Nursing Students' Patient Safety Competencies and Satisfaction With Education Method
Brief Title: Patient Safety Training With The Reverse Face Training Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Vildan Budak, Research Assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Eastern EMU
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Nursing Student; Flipped Education Model
Keywords: nursing student,; patient safety,; flipped education model,; nursing education

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Educational Model (Experimental): Giving the subject of patient safety education with the flipped education model
  Interventions: Other: patient safety competency; Other: satisfaction with the training method
- Traditional Educatıonal Model (Active Comparator): Giving the subject of patient safety education with the traditional education model
  Interventions: Other: patient safety competency; Other: satisfaction with the training method

INTERVENTIONS:
Other: patient safety competency — Investigation of the effect of patient safety education given with the flipped education model and traditional education model on the competence levels of the students.
Other: satisfaction with the training method — Investigation of the effect of patient safety education given with the flipped education model and traditional education model on the satisfaction levels of the students from the education methods.

SUMMARY:
Patient safety is one of the indispensable parts of nursing education. Educating future healthcare professionals about patient safety is very important in terms of providing safe and quality service. In order to include patient safety in the education of nursing students and to determine the effectiveness of the education given, it is necessary to regularly evaluate their knowledge, skills and attitudes about patient safety. At this point, this study was planned in order to increase the awareness of senior nursing students about patient safety before graduation, to evaluate their knowledge, skills and attitudes, to improve the quality of patient care after graduation, and to help minimize or eliminate the possibility of making medical errors. The aim of this study is to examine the effect of the flipped education model on the patient safety competencies of nursing students and their satisfaction with the education method.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines patient safety as "the absence of preventable harm in the health care process and minimizing the unnecessary risks associated with health care service" . In addition, patient safety is the primary and indispensable condition of quality and qualified health services, and it refers to the avoidance of medical errors at every stage of health care by health institutions and employees in the institution and all the precautions taken in order to prevent the harm that health care services may cause to individuals. However, WHO reports that patients encounter many harmful situations while receiving health care services. It has been reported that one out of every ten patients suffers serious damage due to medical errors, and around ten million people are disabled or even lost their lives due to preventable malpractices worldwide every year. It is stated that the most common medical errors are related to drug administration, misuse of equipment and biological accidents. In studies conducted in the United States, it is emphasized that the number of deaths due to medical errors is higher than the number of deaths from traffic accidents, breast cancer or AIDS, and it is stated that medical errors that directly affect patient safety are ranked fifth among the causes of death. In Turkey, it has been reported that official records on patient safety are available to a limited extent, although many people die or become disabled due to medical errors each year. This situation further reveals the importance of the concept of patient safety.

Nurses, who serve their patients 24/7 in hospitals, work actively in all areas, can make quick decisions and think critically, have a key role in ensuring and maintaining patient safety. In order to actively ensure patient safety, nurses need to develop their knowledge, attitudes, skills and competencies regarding patient safety. At this point, the education that nurses have received since their student years is of great importance. During their education, student nurses are tried to gain theoretical and psychomotor skills with a traditional approach in classrooms, laboratory environments and clinics. However, due to the increasing number of students, lack of laboratory conditions, time constraints, and lack of teaching staff, the development of knowledge and skills of nursing students may be insufficient. Students who go to clinical practice before the desired level of knowledge and skill development is completed may encounter the situation of making medical mistakes for the first time, as they experience the anxiety of intervening with the real patient other than the model/mannequin, and also the anxiety of taking notes. In addition, they may witness medical malpractices during clinical practices. In the face of these situations that threaten patient safety, it is recommended that different education and training techniques should be applied in order for students to gain the correct knowledge, skills and attitudes, namely competency regarding patient safety. Because today, traditional learning methods are no longer sufficient to attract the attention of students. For this reason, in recent years, the flipped education model has been used together with the traditional education model in nursing education. The flipped education model is a model that covers different teaching methods and is effective on the academic success of students. Flipped education model; It is an innovative learning model blended as information and technology, supported by pre-class and in-class activities.In the flipped education model, the instructor shares the educational materials such as presentations and videos that he has prepared before the lesson with the student, and the students are required to come to the lesson by studying. It enables students to improve their knowledge and skills through activities such as group discussions, case presentations, and brainstorming. In the flipped education model, the instructor prepares the educational materials in line with the needs of the student, and in this education model, the student can study the educational materials personally at any time and place in a flexible time frame before coming to the lesson. In the flipped education model, the student actively participates in the lesson by using learning methods, while the instructor acts as a consultant and differs from the traditional learning model in these aspects. When the studies on the flipped education model and patient safety competency are examined in the literature; Kim et al. reported a significant increase in patient safety competency between pretest and posttest results in the study titled "The effects of a patient safety course using the flipped classroom approach among nursing undergraduate students: A quasi-experimental study". In other words, they stated that flipped education increases the patient safety knowledge, skills and attitudes of nursing students. Cho et al reported that simultaneous online patient safety education improved the knowledge and skills of nursing students in their study titled "The effect of online education on knowledge, attitudes and skills of nursing students in Korea: a mixed method study" . Torkaman et al. reported that patient safety education is partially effective in improving the patient safety competencies of nursing students in their study titled "The Effect of Patient Safety Education on the Patient Safety Competencies of Nursing Undergraduate Students". Fırat Kılıç and Cevheroğlu , in their study titled "Patient Safety Competencies of Nursing Students", reported that the knowledge, skills and attitudes of nursing students on patient safety were satisfactory and that the students got the lowest score from the patient safety competency scale in the knowledge sub-dimension. Huang et al. in their study "Self-reported confidence in patient safety competencies among Chinese nursing students: a multisite cross-sectional survey" stated that fourth-year nursing students had moderate patient safety competencies.

In conclusion, patient safety is one of the indispensable parts of nursing education. Educating future healthcare professionals about patient safety is very important in terms of providing safe and quality service. In order to include patient safety in the education of nursing students and to determine the effectiveness of the education given, it is necessary to regularly evaluate their knowledge, skills and attitudes about patient safety. At this point, this study was planned in order to increase the awareness of senior nursing students about patient safety before graduation, to evaluate their knowledge, skills and attitudes, to improve the quality of patient care after graduation, and to help minimize or eliminate the possibility of making medical errors. The aim of this study is to examine the effect of the flipped education model on the patient safety competencies of nursing students and their satisfaction with the education method.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th year student at Eastern Mediterranean University, Faculty of Health Sciences, Department of Nursing
* Volunteering to participate in the study,
* Studying in the Turkish department

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
The effect of patient safety training given with the flipped training model on patient safety competence | 6 weeks
  Patient safety competence scale will be used before and after patient safety training, which will be given with flipped training. The scale has a multidimensional structure, consisting of 3 dimensions, 12 factors and a total of 41 items. Item total score averages are used in the total scale and sub-dimensions. The minimum score that can be obtained from the scale and its sub-dimensions is 1 and the maximum score is 5. Items 38 and 39 of the scale are reverse items and should be reverse scored in the evaluation. Higher mean scores indicate that students have better knowledge, skills and attitude competencies regarding patient safety. Permission to use the scale was received by the author via e-mail.
The effect of the patient safety training given with the flipped training model on the level of satisfaction | 6 weeks
  After the patient safety training, which will be given with the flipped training model, a satisfaction survey will be used from the training method.The survey consists of 16 propositions. One of these propositions is the proposition "In general, I am satisfied with this education method", which questions the level of satisfaction with education. Other propositions are generally composed of propositions that aim to determine the student's views on the contribution of the education method to the student's learning and professional life. It is determined that as the scale score increases, students' satisfaction with the education method increases, and as the average scale score decreases, their satisfaction with the education method decreases. In the evaluation of the scale, a minimum of 16 and a maximum of 80 points are given for students' satisfaction with educational methods. Permission to use the scale was received by the author via e-mail.
The effect of patient safety education given with the traditional education model on patient safety competence | 6 weeks
  The patient safety competence scale will be used before and after the patient safety:training, which will be given with the traditional training model. Item total score averages are used in the total scale and sub-dimensions. The minimum score that can be obtained from the scale and its sub-dimensions is 1 and the maximum score is 5. Items 38 and 39 of the scale are reverse items and should be reverse scored in the evaluation. Higher mean scores indicate that students have better knowledge, skills and attitude competencies regarding patient safety. Since the tool is a multidimensional scale, the scale total, 3 dimensions and the score averages of the 12 factors are evaluated separately. Permission to use the scale was received by the author via e-mail.
The effect of patient safety education given with the traditional education model on the level of satisfaction | 6 weeks
  A satisfaction survey will be used from the training method after the patient safety training, which will be given with the traditional training model.The survey consists of 16 propositions. One of these propositions is the proposition "In general, I am satisfied with this education method", which questions the level of satisfaction with education. Other propositions are generally composed of propositions that aim to determine the student's views on the contribution of the education method to the student's learning and professional life. It is determined that as the scale score increases, students' satisfaction with the education method increases, and as the average scale score decreases, their satisfaction with the education method decreases. In the evaluation of the scale, a minimum of 16 and a maximum of 80 points are given for students' satisfaction with educational methods. Permission to use the scale was received by the author via e-mail.

CONTACTS AND LOCATIONS:
Overall Officials: Hülya F Kılıç, Assoc. Prof, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No
will be re-evaluated at the end of the study.

REFERENCES:
- [Result] Stone R, Cooke M, Mitchell M. Undergraduate nursing students' use of video technology in developing confidence in clinical skills for practice: A systematic integrative literature review. Nurse Educ Today. 2020 Jan;84:104230. doi: 10.1016/j.nedt.2019.104230. Epub 2019 Oct 23. PMID 31689584
- [Result] Eskici GT, Kanig M, Ugur E, Seren AKH. The Turkish version of the Patient Safety Competency Self-Evaluation Tool: A validity and reliability study. Nurse Educ Pract. 2021 Nov;57:103229. doi: 10.1016/j.nepr.2021.103229. Epub 2021 Oct 13. PMID 34673387
- [Result] Gurpinar E, Alimoglu MK, Mamakli S, Aktekin M. Can learning style predict student satisfaction with different instruction methods and academic achievement in medical education? Adv Physiol Educ. 2010 Dec;34(4):192-6. doi: 10.1152/advan.00075.2010. PMID 21098386
- [Result] Svitlica BB, Sajnovic M, Simin D, Ivetic J, Milutinovic D. Patient safety: Knowledge and attitudes of medical and nursing students: Cross-sectional study. Nurse Educ Pract. 2021 May;53:103089. doi: 10.1016/j.nepr.2021.103089. Epub 2021 May 18. PMID 34049090
- [Result] Huang FF, Shen XY, Chen XL, He LP, Huang SF, Li JX. Self-reported confidence in patient safety competencies among Chinese nursing students: a multi-site cross-sectional survey. BMC Med Educ. 2020 Jan 31;20(1):32. doi: 10.1186/s12909-020-1945-8. PMID 32005224
- [Result] Firat Kilic H, Cevheroglu S. Patient safety competencies of nursing students. Nurse Educ Today. 2023 Feb;121:105666. doi: 10.1016/j.nedt.2022.105666. Epub 2022 Nov 29. PMID 36463791
- [Result] Torkaman M, Sabzi A, Farokhzadian J. The Effect of Patient Safety Education on Undergraduate Nursing Students' Patient Safety Competencies. Community Health Equity Res Policy. 2022 Jan;42(2):219-224. doi: 10.1177/0272684X20974214. Epub 2020 Nov 26. PMID 33241983
- [Result] Cho DB, Lee W, Kim SY, Choi S. Effect of online education on the knowledge on, attitudes towards, and skills in patient safety for nursing students in Korea: a mixed-methods study. J Educ Eval Health Prof. 2022;19:14. doi: 10.3352/jeehp.2022.19.14. Epub 2022 Jun 30. PMID 35918141
- [Result] Kim YM, Yoon YS, Hong HC, Min A. Effects of a patient safety course using a flipped classroom approach among undergraduate nursing students: A quasi-experimental study. Nurse Educ Today. 2019 Aug;79:180-187. doi: 10.1016/j.nedt.2019.05.033. Epub 2019 May 23. PMID 31153088
- [Result] Park I, Suh Y. Meta-Analysis of Flipped Learning Effects in Nursing Education. Int J Environ Res Public Health. 2021 Dec 5;18(23):12814. doi: 10.3390/ijerph182312814. PMID 34886540
- [Derived] Budak V, Kilic HF, Cevheroglu S. The Impact of a Flipped Learning on Nursing Students' Patient Safety Competencies and Satisfaction With the Education Method: A Randomized Controlled Trial. Nurs Health Sci. 2025 Mar;27(1):e70068. doi: 10.1111/nhs.70068. PMID 40012009